CLINICAL TRIAL: NCT05991661
Title: A Randomized, Double-blind, Placebo-controlled, Multiple Ascending Dose Phase Ib Clinical Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of XKH001 Injection in Healthy Subjects
Brief Title: XKH001 Injection in Healthy Subjects
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Beijing Kanova Biopharmaceutical Co., LTD (Industry)
Responsible Party: Sponsor
Organization: Zhejiang Kanova Biopharmaceutical Co., LTD (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: XKH001-102
Record Dates: First submitted 2023-07-24; First posted 2023-08-14 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-03

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- XKH001 Injection (Active Comparator): Cohort 1: 100 mg Q4W (D1, D29, D57) 6subjects Cohort 2: 300 mg Q4W (D1, D29, D57) 6subjects Cohort 3: 600 mg Q4W (D1, D29, D57) 6subjects The Sponsor will discuss with the investigator to decide whether to conduct the 4th to 5th cohorts (e.g., 600 mg Q14D, 600 mg Q8W, and the specific dose regimen will be determined at that time) no later than the completion of the safety assessment for Cohort 3.
  Interventions: Drug: XKH001 Injection
- XKH001 Placebo Injection (Placebo Comparator): Cohort 1: 100 mg Q4W (D1, D29, D57) 6subjects Cohort 2: 300 mg Q4W (D1, D29, D57) 6subjects Cohort 3: 600 mg Q4W (D1, D29, D57) 6subjects The Sponsor will discuss with the investigator to decide whether to conduct the 4th to 5th cohorts (e.g., 600 mg Q14D, 600 mg Q8W, and the specific dose regimen will be determined at that time) no later than the completion of the safety assessment for Cohort 3.
  Interventions: Drug: XKH001 Placebo Injection

INTERVENTIONS:
Drug: XKH001 Injection — 100mg/ml，1ml/vial
  Other Names: XKH001
  Arms: XKH001 Injection
Drug: XKH001 Placebo Injection — 1ml/vial
  Other Names: XKH001 Placebo
  Arms: XKH001 Placebo Injection

SUMMARY:
This study is a randomized, double-blind, placebo-controlled, multiple ascending dose (MAD) clinical study. The primary objective is to evaluate the safety, tolerability, and PK of multiple SC doses of XKH001 in healthy subjects.

DETAILED DESCRIPTION:
A total of 5 cohorts are planned, with 8 subjects (6 on XKH001 and 2 on placebo) in each cohort. The dosing schedule for the first 3 cohorts is as follows:

Cohort Dosing Regimen

1. 100 mg Q4W (D1, D29, D57)
2. 300 mg Q4W (D1, D29, D57)
3. 600 mg Q4W (D1, D29, D57) After completion of a 6-week safety observation (D1~D43) in the previous cohort, the safety data will be reviewed (blinded) by the investigator and the Sponsor to assess the safety and tolerability of the investigational product. If the dose regimen for the previous cohort is confirmed to be safe and tolerable, dose escalation will continue to the next cohort.

The Sponsor will discuss with the investigator to decide whether to conduct the 4th to 5th cohorts (e.g., 600 mg Q14D, and the specific dose regimen will be determined at that time) no later than the completion of the safety assessment for Cohort 3.

Healthy subjects will be screened within 7 days prior to the first dose and successfully screened subjects will be assigned to the currently ongoing cohort and randomized to receive XKH001 or placebo. Subjects will be admitted to the study site the day before each scheduled dose (D-1, or D28, or D56), complete necessary pre-dose safety assessments, receive SC injection of XKH001 or placebo on D1, or D29, or D57, respectively, and continue to undergo regular safety assessment procedures and other blood sampling (PK, PD, and ADA) after dosing.

Subjects will also undergo comprehensive safety assessments on D15, D43, D71, D85, D113, D141 and D169, including AEs/serious adverse events (SAEs), vital signs, physical examinations, laboratory tests (hematology, blood chemistry, coagulation, urinalysis), 12-lead ECG, etc. Safety data as of D43 will be used by the Sponsor and investigator to assess the safety and tolerability of the investigational product.

If a subject discontinues treatment prematurely, the "Early Withdrawal" visit and all procedures will be performed as on D169.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects who voluntarily sign a written informed consent form (ICF) and are able to complete the study as required by the protocol;
2. Male or female subjects aged 18 to 65 years (inclusive);
3. Subjects with BMI between 18 and 28 kg/m2 (inclusive);
4. Subjects with normal or abnormal but not clinically significant results of vital signs, physical examinations, laboratory tests, 12-lead ECGs and QTcF ≤ 450 ms;
5. Subjects who did not use any prescription or over-the-counter medications within two weeks prior to dosing;
6. Subjects who agree to have no child-bearing plans and to voluntarily take effective contraception measures during the study and within 6 months after the end of the study.

Exclusion Criteria:

1. Pregnant or lactating women;
2. Subjects with clinically significant diseases that may affect the subject's participation in this study within 5 years as judged by the investigator: including but not limited to gastrointestinal, renal, liver, lung, neurological, blood, endocrine, tumor, metabolic, psychiatric or cardio-cerebrovascular diseases, etc.;
3. Subjects with history of autoimmune diseases, known family history of inherited immunodeficiency disorders, or recurrent infections suggestive of possible immunodeficiency;
4. Subjects with active infections requiring hospitalization or IV antibiotic treatment within 3 months prior to dosing, or bacterial, viral and fungal infections with clinical symptoms within 1 week;
5. Subjects with a history of active tuberculosis or subjects with active or latent tuberculosis infection at screening;
6. Subjects with positive HBsAg in 5 items of hepatitis B serology (if HBsAg is negative, HBcAb is positive, and HBsAb is negative, HBV DNA quantitative test is required to be performed [the subject will be excluded if the test result is positive]), positive hepatitis C antibody, treponema pallidum antibody, HIV antigen/antibody;
7. Subjects who plan to receive live or live attenuated vaccines within 4 weeks prior to dosing or during the study;
8. Subjects who have participated in clinical studies of any drug or device within 3 months or 5 half-lives of the investigational product (whichever is longer) prior to dosing;
9. Subjects who are allergic to the investigational product or any component of the formulation of the investigational product or have a history of allergy to protein drugs;
10. Subjects who have consumed more than 14 units of alcohol per week (1 unit of alcohol = 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 6 weeks prior to screening or have taken alcoholic products 1 day before dosing;
11. Subjects who have a history of abuse of other drugs within 5 years prior to screening, or who have a positive urine drug screen result;
12. Subjects who have a smoking history (> 5 cigarettes/day) within 3 months prior to screening;
13. Subjects who have blood donation or blood loss of more than 450 mL within 8 weeks prior to screening, or blood donation of more than 200 mL or blood loss of more than 300 mL within 1 month;
14. Subjects with obstructed venous access or intolerance to venipuncture;
15. Subjects who are considered inappropriate for the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2023-12-01 (Estimated); Primary Completion 2024-08-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AEs) and serious adverse events (SAEs); | From baseline to 24 weeks of follow-up
  Incidence of adverse events (AEs) and serious adverse events (SAEs);
laboratory tests 1 | From baseline to 24 weeks of follow-up
  general condition
laboratory tests 2 | From baseline to 24 weeks of follow-up
  skin and mucosa
laboratory tests 3 | From baseline to 24 weeks of follow-up
  lymph nodes
laboratory tests 4 | From baseline to 24 weeks of follow-up
  head
laboratory tests 5 | From baseline to 24 weeks of follow-up
  neck
laboratory tests 6 | From baseline to 24 weeks of follow-up
  chest
laboratory tests 7 | From baseline to 24 weeks of follow-up
  abdomen
laboratory tests 8 | From baseline to 24 weeks of follow-up
  spine/extremities
observation of injection site | 2 h (± 30 min) post-dose and 4 h (± 30 min) post-dose
  The specific time of observation of injection site reactions is 2 h (± 30 min) post-dose and 4 h (± 30 min) post-dose.
Vital signs | From baseline to 24 weeks of follow-up
  Vital signs include temperature, pulse, and blood pressure. Vital signs will be measured within 60 min before dosing, 2 h (± 30 min), 4 h (± 30 min) after dosing on each dosing day (D1, or D29, or D57); at other visits, vital signs should be measured once.
Hematology | From baseline to 24 weeks of follow-up
  Hematology should include hemoglobin, red blood cell (RBC) count, mean corpuscular hemoglobin, mean corpuscular volume, platelet count, white blood cell (WBC) count, and absolute and percentage of NEUT, LYM, and EOS.
Blood chemistry | From baseline to 24 weeks of follow-up
  Blood chemistry should include fasting glucose, total cholesterol, low-density lipoprotein, high-density lipoprotein, triglycerides, total protein, albumin, aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), lactate dehydrogenase, total bilirubin, direct bilirubin, indirect bilirubin, gamma-glutamyl transpeptidase, creatinine, urea, sodium, potassium, calcium, inorganic phosphorus, chloride, serum lipase, and serum amylase.
Hematology includes: activated partial thromboplastin time (APTT), international normalized ratio (INR), and prothrombin time (PT). | From baseline to 24 weeks of follow-up
  Hematology includes: activated partial thromboplastin time (APTT), international normalized ratio (INR), and prothrombin time (PT).
Three items of thyroid function | From baseline to 24 weeks of follow-up
  Three items of thyroid function should include: FT3, FT4 and TSH.
Urinalysis | From baseline to 24 weeks of follow-up
  Urinalysis should include specific gravity, potential of hydrogen (pH), glucose, bilirubin, urobilinogen, protein, ketones, and occult blood.
12-lead ECGs | From baseline to 24 weeks of follow-up
  12-lead ECGs will be performed at screening, 60 min (± 10 min), 30 min (± 10 min), 15 min (± 10 min) pre-dose on D1, 4 h (± 30 min) post-dose on D1, 4 h (± 30 min) post-dose on D15, D28, and D29, 4 h (± 30 min) post-dose on D43, D56, and D57, and on D58 (approximately 24 h), D59 (approximately 48 h), D61 (approximately 96 h), D64 (approximately 168 h), D71 (approximately 336 h), D85 (approximately 672 h), D113 (approximately 1344 h), D141 (approximately 2016 h), and D169 (approximately 2688 h); before dosing on D1, 3 ECGs should be obtained each time, with an interval of 1-2 min. ECGs from D58 to D169 should be completed within 10 min before PK blood sampling at the current visit for 3 consecutive times, with an interval of approximately 1-2 min.
Infectious disease | From baseline to 24 weeks of follow-up
  Infectious disease testing should include 5 items of hepatitis B serology (hepatitis B surface antigen, hepatitis B surface antibody, hepatitis B e antigen, hepatitis B e antibody, hepatitis B core antibody), hepatitis C antibody, treponema pallidum antibody, and HIV antigen/antibody. If the subject is negative for HBsAg, positive for HBcAb, and negative for HBsAb, HBV DNA testing is also required.
Anteroposterior chest X-ray | From baseline to 24 weeks of follow-up
  Anteroposterior chest X-ray obtained within 3 months before screening is acceptable, and abdominal color ultrasonography obtained within 1 month before screening is acceptable.
PK Cmax | From baseline to 24 weeks of follow-up
  Cmax,ss（Maximum observed concentration）
PK Cmin | From baseline to 24 weeks of follow-up
  Cmin,ss（Minimum observed concentration）
PK Cavg | From baseline to 24 weeks of follow-up
  Cavg,ss（Mean observed concentration）
PK AUC0-inf | From baseline to 24 weeks of follow-up
  AUC0-inf,ss（Area under the serum concentration-time curve from zero to infinity）
PK AUC0-t | From baseline to 24 weeks of follow-up
  AUC0-t,ss（Area under the serum concentration-time curve from zero to t）
PK Tmax | From baseline to 24 weeks of follow-up
  Tmax,ss（Time of observed）
PK t1/2 | From baseline to 24 weeks of follow-up
  t1/2,ss（Terminal half-life）
PK AUCtau | From baseline to 24 weeks of follow-up
  area under the serum concentration-time curve at steady state (AUCtau)
PK %AUCex | From baseline to 24 weeks of follow-up
  percentage of extrapolated area under the serum concentration-time curve from zero to infinity at steady state (%AUCex)
PK λz | From baseline to 24 weeks of follow-up
  elimination rate constant of serum concentration in the terminal phase (λz,ss)
PK Rac | From baseline to 24 weeks of follow-up
  drug accumulation ratio (Rac)
PK Vz | From baseline to 24 weeks of follow-up
  volume of distribution at steady state (Vz,ss/F)
PK CL | From baseline to 24 weeks of follow-up
  clearance at steady state (CLss/F)
PK MRT | From baseline to 24 weeks of follow-up
  mean residence time (MRT)

SECONDARY OUTCOMES:
Total IgE; | From baseline to 24 weeks of follow-up
  Total Immunoglobulin E（IgE）;
EOS count in whole blood; | From baseline to 24 weeks of follow-up
  Eosinophil（EOS） count in whole blood;
NEUT count in whole blood; | From baseline to 24 weeks of follow-up
  Neutrophil（NEUT） count in whole blood;
Blood LYM count; | From baseline to 24 weeks of follow-up
  Blood Lymphocyte(LYM) count;
Levels of IL-25-related cytokines in serum | From baseline to 24 weeks of follow-up
  Levels of IL-25-related cytokines in serum (multiple cytokine panel includes: IL-25, TARC, IL-8, MIP1β, Eotaxin, CXCL1 (KC/GROα), Eotaxin-3);
ADA | From baseline to 24 weeks of follow-up
  Incidence of anti-drug antibodies (ADAs).

OTHER OUTCOMES:
QT/QTc | From baseline to 24 weeks of follow-up
  Relationship between multiple-dose serum concentrations and QTcF

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, Principal Investigator — The First Hospital of Jilin University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang H, Zheng W, Peng R, Wu D, Hu Y, Sun T, Gao L, Liu Y, Guo L, Ding Y, Liu L. First-in-human study on tolerability, pharmacokinetics and pharmacodynamics of single and multiple escalating doses of XKH001, a recombinant humanized monoclonal antibody against IL-25 in healthy Chinese volunteers. Expert Opin Investig Drugs. 2025 Jan-Feb;34(1-2):81-87. doi: 10.1080/13543784.2025.2453162. Epub 2025 Jan 20. PMID 39815604